CLINICAL TRIAL: NCT05090319
Title: Use of a Micro-hematology Analyzer for Discriminating Between Viral and Bacterial Infections in Hospitalized Adults: An Observational Study
Brief Title: Micro-hematology Analyzer for Viral/Bacterial Description
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RizLab Health, Inc. (Industry)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: H-49795
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Infection Viral; Infection, Bacterial
MeSH Terms: conditions — Virus Diseases; Bacterial Infections | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Viral Group: known viral infection
  Interventions: Diagnostic Test: complete blood count
- Bacterial group: known bacterial infection
  Interventions: Diagnostic Test: complete blood count

INTERVENTIONS:
Diagnostic Test: complete blood count — Complete blood count will be performed on the patient. Accuracy of micro-hematology analyzer will be assessed.

SUMMARY:
The purpose of the study is to evaluate the reliability and accuracy of a newly developed point-of-care analyzer, theCytoTracker, to measure complete blood count (CBC) parameters and discriminate between viral and bacterial infections.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the reliability and accuracy of a newly developed point-of-care analyzer, the CytoTracker, to measure complete blood count (CBC) parameters. The CytoTracker results will be compared to those from a standard benchtop analyzer (Horiba Point of Care Hematology Analyzer, ABX Micros ES 60). If successful, the data from this study would be used to support a pre-submission meeting to the FDA for the CytoTracker. In addition to validating the CytoTracker, the project will study the use of CBC parameters to distinguish between observed bacterial or viral infections in adults. Hospitalized adult subjects with suspected or confirmed viral or bacterial infections will be enrolled in the study. After enrollment a venous blood sample (baseline sample) will be collected and the CytoTracker will be used to measure CBC parameters (cell counts and population distribution). Clinical data will be abstracted from the medical record and used with the CBC parameters to develop an algorithm to distinguish between bacterial and viral infections.

ELIGIBILITY:
Inclusion Criteria:

-COVID positive or suspected/confirmed bacterial infection (lower UTI, pneumonia, septecemia, etc). -Adults 18 years of age and older. -Meet SIRS criteria anytime during the ED presentation.

Exclusion Criteria:

* Subjects who are unable to give informed consent will be excluded
* Subjects with the following conditions will also be excluded: Known white blood cell, neutrophil, and lymphocyte disorders Active cancer patients; For solid tumors, subject will be excluded if he/she has received chemotherapy in the last 3 months.
* Subjects who are pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Emergency room patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-07-24 (Estimated); Study Completion 2022-07-24 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 1 year
  Accuracy of Device in quantifying WBC, Neutrophils, and Lymphocytes; Accuracy of Viral/Bacterial Descrimination

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller J, Starks B. Deciphering clues in the CBC count. Nursing. 2010 Jul;40(7):52-5. doi: 10.1097/01.NURSE.0000383454.33035.4b. No abstract available. PMID 20548208
- [Background] Korppi M, Kroger L, Laitinen M. White blood cell and differential counts in acute respiratory viral and bacterial infections in children. Scand J Infect Dis. 1993;25(4):435-40. doi: 10.3109/00365549309008524. PMID 8248742
- [Background] Juul S, Pliskin JS, Fineberg HV. Variation and information in white blood cell differential counts. Med Decis Making. 1984;4(1):69-80. doi: 10.1177/0272989X8400400110. PMID 6727589
- [Background] Kramer MS, Tange SM, Mills EL, Ciampi A, Bernstein ML, Drummond KN. Role of the complete blood count in detecting occult focal bacterial infection in the young febrile child. J Clin Epidemiol. 1993 Apr;46(4):349-57. doi: 10.1016/0895-4356(93)90149-u. PMID 8482999
- [Background] Jung YJ, Kim JH, Park YJ, Kahng J, Lee H, Lee KY, Kim MY, Han K, Lee W. Evaluation of cell population data on the UniCel DxH 800 Coulter Cellular Analysis system as a screening for viral infection in children. Int J Lab Hematol. 2012 Jun;34(3):283-9. doi: 10.1111/j.1751-553X.2011.01392.x. Epub 2012 Jan 9. PMID 22226427
- [Background] Chaves F, Tierno B, Xu D. Quantitative determination of neutrophil VCS parameters by the Coulter automated hematology analyzer: new and reliable indicators for acute bacterial infection. Am J Clin Pathol. 2005 Sep;124(3):440-4. doi: 10.1309/LLF7-5W0F-WQQ8-TCC5. PMID 16191513
- [Background] Naess A, Nilssen SS, Mo R, Eide GE, Sjursen H. Role of neutrophil to lymphocyte and monocyte to lymphocyte ratios in the diagnosis of bacterial infection in patients with fever. Infection. 2017 Jun;45(3):299-307. doi: 10.1007/s15010-016-0972-1. Epub 2016 Dec 19. PMID 27995553
- [Background] Furniturewalla A, Chan M, Sui J, Ahuja K, Javanmard M. Fully integrated wearable impedance cytometry platform on flexible circuit board with online smartphone readout. Microsyst Nanoeng. 2018 Jul 30;4:20. doi: 10.1038/s41378-018-0019-0. eCollection 2018. PMID 31057908
- [Background] Ahuja K, Rather GM, Lin Z, Sui J, Xie P, Le T, Bertino JR, Javanmard M. Toward point-of-care assessment of patient response: a portable tool for rapidly assessing cancer drug efficacy using multifrequency impedance cytometry and supervised machine learning. Microsyst Nanoeng. 2019 Jul 15;5:34. doi: 10.1038/s41378-019-0073-2. eCollection 2019. PMID 31645995
- [Background] Power M, Fell G, Wright M. Principles for high-quality, high-value testing. Evid Based Med. 2013 Feb;18(1):5-10. doi: 10.1136/eb-2012-100645. Epub 2012 Jun 27. PMID 22740357